CLINICAL TRIAL: NCT04535674
Title: A Multicenter, Randomised, Controlled, Open Label Trial on the Efficacy and Safety of Asunercept for Patients With Severe COVID-19 Disease
Brief Title: Asunercept in Patients With Severe COVID-19
Acronym: ASUNCTIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apogenix AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APG101_CD_017; 2020-001887-27 (EudraCT Number)
Record Dates: First submitted 2020-08-31; First posted 2020-09-02 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-07

CONDITIONS: COVID-19 Induced Pneumonia; Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Asunercept/APG101 will be tested in three parallel intervention arms and compared with Standard of Care (SoC). The study will compare treatment efficacy of SoC to that of weekly intravenous infusions of Asunercept at three different doses. Patients will be randomised into four groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard of Care (No Intervention)
- Standard of Care + Asunercept 25 mg (Experimental)
  Interventions: Biological: Asunercept
- Standard of Care + Asunercept 100 mg (Experimental)
  Interventions: Biological: Asunercept
- Standard of Care + Asunercept 400 mg (Experimental)
  Interventions: Biological: Asunercept

INTERVENTIONS:
Biological: Asunercept — Asunercept (APG101) will be administered once per week as an i.v. infusion
  Arms: Standard of Care + Asunercept 100 mg; Standard of Care + Asunercept 25 mg; Standard of Care + Asunercept 400 mg

SUMMARY:
This is an open-label, randomized, phase II study with the main objective to investigate the effectiveness and safety of an investigational drug (APG101; International Nonproprietary Name: asunercept) in patients with severe COVID-19 disease. The study aims to decrease overall and SARS-CoV-2 associated pneumonia mortality in patients with COVID-19 as well as to decrease the percentage of patients admitted to Intensive Care Unit (ICU), decrease the need to supply oxygen to patients, reduce the number of days patients are hospitalized in ICU and/or on the ward, decrease the number of days required to obtain a negative result in the PCR (Polymerase Chain Reaction, a laboratory technique that allows the amplification of small fragments of DNA to detect the presence of the virus) test for COVID-19 and decrease the levels of markers that indicate pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory confirmed infection with SARS-CoV-2 OR typical radiological signs of SARS-CoV-2 infection
* Hospitalisation due to COVID-19
* Informed Consent obtained, the patient understands and agrees to comply with the planned study procedures. If a potential patient is unconscious, the Patient Information Sheet with the Informed Consent Form can be signed by the legal representative, if he/she accompanies the patient. It can be signed by a Concilium consisting of doctors (2), investigator and an independent witness in case the legal representative is not available.
* ≥18 years of age
* Willingness to perform effective measures of contraception during the study.
* Signs of respiratory deterioration such as oxygen saturation ≤94% when breathing ambient air or >3% drop in oxygen saturation in case of chronic obstructive lung disease OR need for oxygen supplementation to achieve satisfactory blood oxygen saturation (sPO2>90% at room air) as well as the need for non-invasive ventilation, high-flow oxygen devices or mechanical ventilation or radiological or clinical signs of pneumonia.

Exclusion Criteria:

* Moribund, or estimated life expectancy <1 month (e.g., terminal cancer, etc.)
* Patient does not qualify for intensive care, based on local triage criteria
* Pregnancy or breast feeding
* Severe liver dysfunction (e.g. ALT/AST > 5 times upper limit of normal)
* Anticipated discharge from hospital within 48 hours
* Other potent anti-inflammatory treatment, e.g. TNF- blocking therapies
* Mechanical ventilation for >48 hours
* Known active HIV or viral hepatitis infection
* Known active tuberculosis
* Known hereditary fructose intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Time to sustained improvement of one category (i.e. two consecutive days) from randomisation | Day 1-29
  The primary endpoint is time to clinical improvement which is defined as time from randomisation to an (sustained) improvement of at least one category on two consecutive days compared to the status at randomisation measured on a nine-category ordinal scale (proposed by WHO).

SECONDARY OUTCOMES:
Efficacy according to the National Early Warning Score (NEWS) | Day 1-29
  Time to discharge or to a NEWS of ≤2 and maintained for 24 hours, whichever occurs first Change from baseline
Oxygenation | Day 1-29
  Oxygenation free days until day 29 Incidence and duration of new oxygen use during the trial
Ventilation | Day 1-29
  Ventilator free days until day 29 Incidence and duration fo new mechanical ventilation use during the trial
Hospitalisation - Length | Day 1-29
  Duration of hospitalisation Length of ICU stay (in days)
Hospitalisation - Proportion on ICU | Day 1-29
  Proportion of patients admitted to ICU
Mortality | Up to 90 days
  15-day, 29-day, 60-day and 90-day all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Ruiz-Seco, PhD-MD, Principal Investigator — Hospital Universitario Infanta Sofía, Madrid
Locations (13):
- Russia (7):
  - Republican Clinical Infectious Hospital n.a. professor A.F. Agafonov, Kazan'
  - Scientific Research lnstitute fоr Соmрlех lssues of Cardiovascular Diseases, Kemerovo
  - Federal State Budgetary Educational Institution of Higher Education "Kuban State Medical University" of the Ministry of Health of the Russian Federation, Krasnodar
  - State Budgetary Healthcare Institution "Scientific Research Institute - Regional clinical hospital No. 1 n.a. professor S.V. Ochapovsky" of the Ministry of Healthcare of Krasnodar Krai, Krasnodar
  - State Budgetary Institution of Health of the Nizhny Novgorod Region "Infectious Clinical Hospital No. 2 of Nizhny Novgorod", Nizhny Novgorod
  - Ryazan State Medical University n.a. academician I.P. Pavlov, Ryazan
  - Saint Petersburg state budgetary healthcare institution "City hospital of Saint George the great Martyr", Saint Petersburg
- Spain (6):
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Universitario Infanta Sofia, San Sebastián de los Reyes
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruiz Seco MP, Pano Pardo JR, Schoergenhofer C, Dings C, Lehr T, Herth F, Krendyukov A, Straub C, Kappler M, Jilma B, Fricke H, Pardo J, de Miguel D, Thiemann M, Bergmann M, Walczak H, Hoeger T. Efficacy and safety of asunercept, a CD95L-selective inhibitor, in hospitalised patients with moderate-to-severe COVID-19: ASUNCTIS, a multicentre, randomised, open-label, controlled, phase 2 trial. EClinicalMedicine. 2024 Oct 24;77:102879. doi: 10.1016/j.eclinm.2024.102879. eCollection 2024 Nov. PMID 39513186